CLINICAL TRIAL: NCT06377553
Title: PET/MRI Evaluation of Endometriosis Using Intercellular Matrix Radiopharmaceuticals
Brief Title: PET/MRI for Evaluation of Endometriosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Onofrio A. Catalano, MD, PhD, Associate Professor Harvard Medical School, PET/MR Translation Officer, Medical Director PET/MR at the Athinoula A. Martinos Center for Biomedical Imaging, Massachusetts General Hospital
Other Study IDs: 2023P000955
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis; Endometrioma
Keywords: Endometriosis; [18F]-FAPI-74; [68Ga]CBP8-PET; PET/MR; Fibrosis; DIE; Endometrioma
MeSH Terms: conditions — Endometriosis; Fibrosis | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Endometriosis: Patient with clinical diagnosis of endometriosis, in any stage, candidate for diagnostic or therapeutic laparoscopic surgery.
  Interventions: Drug: Radiotracer Injection; Diagnostic Test: Imaging; Other: Rectal Ultrasound Gel Injection

INTERVENTIONS:
Drug: Radiotracer Injection — An intravenous catheter will be placed in an arm or hand vein for injection of [68Ga]CBP8;
  6-10 mCi of [68Ga]CBP8 or 5-9 mCi of FAPI will be injected into the Biograph mMR system. The injected dose and the time of injection will be recorded; The catheter will be flushed with 0.9% saline solution; The subjects will then be positioned on the scanner table; support devices under the back or legs will be used to enable the patient to maintain his/her position throughout the scan comfortably.
Diagnostic Test: Imaging — MRI and PET scanner to be used:
  3.0 T Laboratory (Bay 7) Siemens Biograph mMR.
  Magnetic resonance images of the pelvis and abdomen will be acquired using the Martinos Center's combined 3 Tesla PET/MRI scanner. The image quality on these 3 Tesla devices will be very high, equivalent to or better than any other standard clinical MRI system. PET images of the target body site will be acquired when necessary, the data acquisition will be started shortly before radiotracer injection; Coincidence event data will be acquired and stored in list mode or compressed (i.e., sinogram space) format. Subjects will be asked to lie still for the duration of the study. The entire imaging session will last up to 120 minutes
Other: Rectal Ultrasound Gel Injection — About 50ml of ultrasound gel will be placed into the vagina using the blunt end of the ultrasound gel tube or a Foley catheter or a syringe with a blunt Christmas tree end. No ultrasound probe will be inserted into the vagina, no external ultrasound probe will be used. No ultrasound study will be performed. The ultrasound gel will only be used to distend the vagina and improve the quality of MRI images; this is standard of practice in MRI for endometriosis and for several other gynecological diseases.

SUMMARY:
This study aims to determine if PET/MRI can detect endometriosis and potentially improve upon currently available non-invasive diagnostic capabilities. Specifically, the authors will investigate the ability of PET/MRI to detect and quantify endometriosis, as well as differentiate among subcategories such as inflammatory peritoneal lesions, fibrotic deep infiltrating endometriosis lesions (DIE), and ovarian endometriomas. The authors will compare [68Ga]CBP8 or [18F]-FAPI-74 PET/MRI imaging versus the current gold standard diagnostic methods, including laparoscopic surgery, clinical follow-up, and follow-up imaging.

DETAILED DESCRIPTION:
Several imaging techniques, including ultrasound, computed tomography and magnetic resonance imaging (MRI), have been used for the detection of DIE, for mapping and staging endometriosis. Currently, the modalities most commonly used are transvaginal ultrasound (TVS) and magnetic resonance imaging MRI. TVS is generally considered a first-line technique.TVS, in highly experienced hands, meets the criteria for mapping DIE to the uterosacral ligaments, rectovaginal septum, vaginal wall, pouch of Douglas and rectosigmoid; however it is limited by its operator dependance and by the small field of view (FOV). MRI is commonly used for mapping lesions within the Douglas pouch and rectovaginal septum and rectosigmoid. MRI has shown acceptable diagnostic values, with pooled sensitivity and specificity for pelvic endometriosis of 94% and 77%, respectively. For rectosigmoid endometriosis, MRI's pooled sensitivity and specificity were 92% and 96%, respectively. However, MRI has limitations, specially in the evaluation of chronic fibrotic endometriosis and for assessing the peritoneum and extension beyond the pelvis as well as DIEs. There is a growing body of literature examining the role of PET/MRI in pelvic and abdominal malignancies and its potential superiority to MRI alone. However, there are no studies that used PET/MRI to investigate endometriosis.

This study aims to use [68Ga]CBP8- or [18F]FAPI PET/MRI to diagnose and quantify endometriosis. The novel radiopharmaceutical collagen-binding probe 8 labeled with Gallium-68 selectively binds to collagen type I, the predominant extracellular protein in fibrosis. [68Ga]CBP8 has already been investigated in patients affected by pulmonary fibrosis with success. Fibroblast activation protein (FAP) is a type II transmembrane serine protease that is overexpressed in CAFs and, to a lesser extent, in benign processes. It is associated with extracellular matrix remodeling, for example, chronic inflammation, degenerative bone and spine disease, arthritis, and cardiac remodelling after myocardial infarction. Quinolone-based FAP inhibitors (FAPIs) constitute a class of molecules with high affinity to FAP deployed to assess many types of solid tumors and some benign pathologies. 68Ga-FAPIs and, to a lesser extent, 18F-FAPI are being extensively studied in oncologic and non-oncologic positron emission tomography/computed tomography (PET/CT) and, to a lesser extent, PET/MRI, both in Europe and Asia.

In this single-arm, single-center, open label prospective study, the authors will recruit 60 patients with clinical diagnosis of endometriosis who candidate for laparoscopic surgery. Patients will be referred to FAPI- or CBP8-PET/MRI by their primary treating gynecologist physicians. Laparoscopy will serve as primary standard of reference; clinical and imaging follow up, as well as prior diagnostic imaging studies (CT, MRI, US), will serve as secondary standard of reference. In the case patients will not undergo laparoscopy, then clinical and imaging follow up, as well as prior diagnostic imaging studies (CT, MRI, US), will serve as primary standard of reference.

Board-certified radiologists will evaluate [18F]-FAPI-74 or [68Ga]CBP8-PET/MR images and standalone MR images in a blinded fashion on separate occasions. Assessment of of endometriosis will be performed according to consolidated published criteria for MRI. For endometriosis staging, the readers will follow rASRM criteria. Then, the authors will compare the sensitivity, specificity, and accuracy of regional/whole-body staging using FAPIor CBP-PET/MRI versus regional/wholebody MRI, with the standard reference set as pathology results, when available, or clinical and imaging follow-up otherwise. Hypothesis testing will be performed using McNemar's test for matched pairs testing.

ELIGIBILITY:
Inclusion Criteria:

- Patients with clinical diagnosis of endometriosis, in any stage, candidate for diagnostic overtherapeutic laparoscopic surgery.

Exclusion Criteria:

* Subjects less than 18 years of age or greater than 70 years of age.
* Any contraindication to MRI, including electrical implants, such as cardiac pacemakers or perfusion pumps. MRI non-compatible ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, prosthetic heart valves that are not compatible with the gradient maps of our scanners, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, steel implants, and/or ferromagnetic objects such as jewelry, or metal clips in clothing that cannot be removed.
* History of claustrophobic reactions.
* Individuals who do not speak or understand English since providing a translated version of the entire consent form is not practicable
* Any contraindication to PET including active breastfeeding (a negative STAT quantitative serum hCG pregnancy test is required on the day of the scan before the subject can participate)
* History of research-related radiation exposure exceeding current Radiology Department guidelines (i.e., 50 mSv in the prior 12 months).
* QTc>460msec obtained within 30 days from the PET/MR
* eGFR <60mL/min/1.73m2 obtained within 30 days from the PET/MR
* AST >40U/L and/or ALT >55 U/L obtained within 30 days from the PET/MR
* A greater risk than normal for potential cardiac arrest such as history of non compensated congestive heart failure, poorly controlled arrythmias, symptomatic non compensated cardiopathies.
* History of major head trauma (i.e., multiple concussions, traumatic brain injury).
* History of bleeding disorders.
* Inability to lie comfortably on a bed inside the PET/MRI bore as assessed by physical examination and medical history (e.g., back pain, severe arthritis).
* Subjects under the direct supervision of the principal investigator.
* Body weight of > 300 lbs. (weight limit of the MRI table) or BMI >33.0 per the standard operating procedure of PET/MRI safety at the Martinos Center.
* Subjects from any other at-risk populations (e.g., children and minors cognitively impaired persons, prisoners).

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: In total, 60 subjects with clinically diagnosed endometriosis will be recruited. All subjects recruited for the study will be able to withdraw from the study at any time. The patients will be referred to the study by their treating physicians to investigate clinically diagnosed endometriosis. We will not recruit or enroll healthy volunteers in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-01-03 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of PET/MR in Preoperative Endometriosis Detection | 1-2 Months
  To determine the accuracy, sensitivity, and specificity of [18F]-FAPI-74 and/or [68Ga]CBP8 PET/MRI in detecting and classifying endometriosis, using the gold standard methods as the reference.
Diagnostic Performance of PET/MRI vs. Conventional Imaging | 1-2 Months
  To determine the accuracy, sensitivity, and specificity of [18F]-FAPI-74 or [68Ga]CBP8-PET/MR images versus stand-alone wholebody MRI and/or pelvic MRI and/or ultrasound and/or computed tomography in pre-operative patients with suspected endometriosis lesion.

SECONDARY OUTCOMES:
Impact of [18F]-FAPI-74 and [68Ga]CBP8 PET/MRI on Diagnosis and Management in Endometriosis | 1-6 months
  To determine if imaging with [18F]-FAPI-74 and/or [68Ga]CBP8 PET/MRI results in changes to diagnosis, medical or surgical management in endometriosis patients
Correlation of Pre-Treatment PET Uptake and Post-Treatment Response in Endometriosis | 6-12 months
  To determine if pre-treatment measures of [18F]-FAPI-74 and/or [68Ga]CBP8 standardized uptake values (SUVs) are correlated to post-treatment response in patients with endometriosis.

CONTACTS AND LOCATIONS:
Overall Officials: Onofrio Catalano, Principal Investigator — Athinoula A. Martinos Center for Biomedical Imaging, Massachusetts General Hospital, Harvard Medical School
Locations (1):
- Athinoula A. Martinos Center for Biomedical Imaging, Massachusetts General Hospital, Harvard Medical School, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor HS, Kotlyar AM, Flores VA. Endometriosis is a chronic systemic disease: clinical challenges and novel innovations. Lancet. 2021 Feb 27;397(10276):839-852. doi: 10.1016/S0140-6736(21)00389-5. PMID 33640070
- [Background] Moradi Y, Shams-Beyranvand M, Khateri S, Gharahjeh S, Tehrani S, Varse F, Tiyuri A, Najmi Z. A systematic review on the prevalence of endometriosis in women. Indian J Med Res. 2021 Mar;154(3):446-454. doi: 10.4103/ijmr.IJMR_817_18. PMID 35345070
- [Background] Bazot M, Darai E. Diagnosis of deep endometriosis: clinical examination, ultrasonography, magnetic resonance imaging, and other techniques. Fertil Steril. 2017 Dec;108(6):886-894. doi: 10.1016/j.fertnstert.2017.10.026. PMID 29202963
- [Background] Nisenblat V, Bossuyt PM, Farquhar C, Johnson N, Hull ML. Imaging modalities for the non-invasive diagnosis of endometriosis. Cochrane Database Syst Rev. 2016 Feb 26;2(2):CD009591. doi: 10.1002/14651858.CD009591.pub2. PMID 26919512
- [Background] Saba L, Sulcis R, Melis GB, Ibba G, Alcazar JL, Piga M, Guerriero S. Diagnostic confidence analysis in the magnetic resonance imaging of ovarian and deep endometriosis: comparison with surgical results. Eur Radiol. 2014 Feb;24(2):335-43. doi: 10.1007/s00330-013-3013-9. Epub 2013 Sep 12. PMID 24026621
- [Background] Giesel FL, Adeberg S, Syed M, Lindner T, Jimenez-Franco LD, Mavriopoulou E, Staudinger F, Tonndorf-Martini E, Regnery S, Rieken S, El Shafie R, Rohrich M, Flechsig P, Kluge A, Altmann A, Debus J, Haberkorn U, Kratochwil C. FAPI-74 PET/CT Using Either 18F-AlF or Cold-Kit 68Ga Labeling: Biodistribution, Radiation Dosimetry, and Tumor Delineation in Lung Cancer Patients. J Nucl Med. 2021 Feb;62(2):201-207. doi: 10.2967/jnumed.120.245084. Epub 2020 Jun 26. PMID 32591493
- [Background] Hamson EJ, Keane FM, Tholen S, Schilling O, Gorrell MD. Understanding fibroblast activation protein (FAP): substrates, activities, expression and targeting for cancer therapy. Proteomics Clin Appl. 2014 Jun;8(5-6):454-63. doi: 10.1002/prca.201300095. Epub 2014 Mar 24. PMID 24470260
- [Background] Desogere P, Tapias LF, Hariri LP, Rotile NJ, Rietz TA, Probst CK, Blasi F, Day H, Mino-Kenudson M, Weinreb P, Violette SM, Fuchs BC, Tager AM, Lanuti M, Caravan P. Type I collagen-targeted PET probe for pulmonary fibrosis detection and staging in preclinical models. Sci Transl Med. 2017 Apr 5;9(384):eaaf4696. doi: 10.1126/scitranslmed.aaf4696. PMID 28381537
- [Background] Giesel FL, Kratochwil C, Lindner T, Marschalek MM, Loktev A, Lehnert W, Debus J, Jager D, Flechsig P, Altmann A, Mier W, Haberkorn U. 68Ga-FAPI PET/CT: Biodistribution and Preliminary Dosimetry Estimate of 2 DOTA-Containing FAP-Targeting Agents in Patients with Various Cancers. J Nucl Med. 2019 Mar;60(3):386-392. doi: 10.2967/jnumed.118.215913. Epub 2018 Aug 2. PMID 30072500